CLINICAL TRIAL: NCT06583434
Title: Effects of Stabilization-based Pilates Exercise on Gait and Balance in Women With Flexible Pesplanus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hyun Ju Kim (Other)
Responsible Party: Sponsor-Investigator, Hyun Ju Kim, Principal Investigator, Busan University of Foreign Studies
Organization: Busan University of Foreign Studies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUFS-FF-2023
Record Dates: First submitted 2024-08-29; First posted 2024-09-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Flexible Flatfoot
Keywords: flexible flatfoot; balance; gait; Pilates; pesplanus
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates-Training Group (Experimental): Participants in this group will receive twice-weekly Pilates sessions focusing on core and lower extremity stabilization exercises. Each session will last for 50 minutes and the intervention will continue for 8 weeks. The goal of this intervention is to improve gait patterns and balance in women with flexible flatfoot.
  Interventions: Behavioral: core-lower extremity Pilates Training Group
- Non-Training Group (Experimental): Participants in this group will not receive any specific intervention during the study period. They will continue their usual activities without any additional exercises provided by the study
  Interventions: Other: Non-Training Group

INTERVENTIONS:
Behavioral: core-lower extremity Pilates Training Group — Participants in this group will engage in a stabilization-based Pilates exercise program focusing on core and lower extremity stabilization. The program consists of twice-weekly sessions, each lasting 50 minutes, over a period of 8 weeks. The primary goal of the intervention is to improve gait patterns and balance in women with flexible pes planus
  Arms: Pilates-Training Group
Other: Non-Training Group — Participants in this group will not receive any specific intervention during the study period. They will continue their usual activities without any additional exercises provided by the study.
  Arms: Non-Training Group

SUMMARY:
The goal of this clinical trial was to determine if stabilization-based Pilates exercises could improve gait and balance in women with flexible flatfoot.

The main questions it aimed to answer were:

Did Pilates training improve gait parameters in women with flexible flatfoot? Did Pilates training reduce balance instability in these participants?

Researchers compared the Pilates training group to a non-training group. The results showed significant improvements in gait and balance for those who participated in the Pilates training.

Participants:

Completed twice-weekly Pilates sessions for 8 weeks. Underwent pre- and post-intervention assessments of gait and balance.

DETAILED DESCRIPTION:
Study object This randomized controlled trial aims to assess the effects of stabilization-based Pilates exercises on gait and balance in women with flexible flatfoot. The study focuses on determining whether a specific Pilates program can provide non-invasive rehabilitation for improving gait patterns and reducing balance instability.

Participants The study will include 22 healthy women with flexible flatfoot who have no congenital deformities or diseases of the feet, knees and have a navicular drop of ≥10 mm. The participants will be recruited from "Clinical Pilates" studio in Busan city. Women with bilateral flatfoot (n=22) will be randomly allocated to either the Pilates training group (PTG, n=11) or the non-training group (NTG, n=11).

Outcome measure gait assessment and data acquisition: Participants undergo several practice walks to familiarize themselves with the gait assessment. Three records are averaged once they show a normal gait pattern. The assessment uses measurements from both legs and is conducted in a non-distracting environment.

Seven 3D infrared motion capture cameras (Vicon camera MX-T20, Oxford Metrics, Oxford, UK) and 16 circular reflective markers (14-mm diameter) are used to acquire the data for the gait assessment. The reflective markers are attached to the anterior superior iliac spine, posterior superior iliac spine, lateral mid-thigh, lateral femoral epicondyle, mid-shin, lateral malleolus, second metatarsus, and heel of both the left and right legs. The height, body weight, and width of knee and ankle joints are measured and entered. Gait analysis includes temporal parameters, such as foot-off, step time, stride time, walking speed, and cadence. Kinematic data are collected using Vicon plug-in gait system (Oxford Metrics) at a sampling frequency of 100 Hz.

balance assessment and data acquisition: The participants are instructed to stand with their arms crossed in front of their chest, with one leg supported and one leg raised with the knee at a 90° angle. Participants hold that standing position for 40 seconds. Three successful attempts are recorded for each participant. Measurements are taken for both legs, and the participants are given sufficient time to rest between each stage of the experiment.

For Center of Pressure (COP) measurement, data from 40 seconds of single leg support on a force platform (AMTI-OR6, Watertown, MA, USA) are utilized. The data are calculated and assessed as time series data. COP sway variability is assessed based on the Root Mean Sqaure (RMS) in Anterior-Posterior (AP) and Medial-Lateral (ML) directions, while AP and ML components of COP velocity and range are also assessed. Kinematic data are collected using the Vicon Plug-in Gait system at a sampling frequency of 100 Hz.

Exercise intervention:

The exercise intervention consists of two sessions each week, for a total of 16 sessions over an 8-week period. Each training session is structured into eight sets, totaling 50 minites. This includes a 5-min warm-up period, followed by 40-min of the main exercise component, and concluding with a 5-min cool-down phase. The Pilates training is supervised by an instructor with 15 years of experience and a professional Pilates certification.

Statistical analysis IBM SPSS Statistics for Windows (version 28.0; IBM Corp., Armonk, N.Y., USA) is used to conduct descriptive statistical analyses, including means and standard deviations. Statistical significance is set at p<0.05.

Differences in mean values between the groups for each temporal parameter will be assessed using independent samples t-tests. Additionally, due to the small sample size, non-parametric tests (Mann-Whitney U test) will be conducted. Furthermore, paired samples t-tests will be used for within-group pre-test and post-test comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral navicular drop of ≥10 mm

Exclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease
* Severe heart conditions (heart failure, myocardial infarction)
* History of knee, ankle or hip injuries within the last 3 months
* Chronic lung disease
* Pregnancy
* Congenital Foot Deformity ( Polydactyly, Syndactyly)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change in step time | Baseline and after 8 weeks
  Step time was measured in seconds using a 3D motion capture system.
Change in stride time | Baseline and after 8 weeks
  Stride time was measured in seconds using a 3D motion capture system.
Change in walking speed | Baseline and after 8 weeks
  Walking speed was measured in meters per second using a 3D motion capture system.
Change in cadence | Baseline and after 8 weeks
  Cadence was measured in steps per minute using a 3D motion capture system.
Change in foot off | Baseline and after 8 weeks
  Foot off was measured as a percentage of the gate cycle using a 3D motion capture system.
Change in balance stability | Baseline and after 8 weeks
  Balance was assessed using a single-leg stance test, measuring the center of pressure(COP) sway in both anterior-posterior (AP) and medial-lateral (ML) directions.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Ju Kim, MSc, Principal Investigator — Department of Sports and Health Convergence
Locations (1):
- Busan University of Foreign Studies, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared via Figshare. The data will include demographic information, raw data from the assessments, and any other relevant data collected during the study.
Supporting Information: SAP
Time Frame: The data will be available immediately after the publication of the study results and will be accessible for at least 5 years
Access Criteria: The data will be openly available via Figshare without the need for a data access request

REFERENCES:
- [Background] Abasiyanik Z, Ertekin O, Kahraman T, Yigit P, Ozakbas S. The effects of Clinical Pilates training on walking, balance, fall risk, respiratory, and cognitive functions in persons with multiple sclerosis: A randomized controlled trial. Explore (NY). 2020 Jan-Feb;16(1):12-20. doi: 10.1016/j.explore.2019.07.010. Epub 2019 Jul 17. PMID 31377306
- [Background] Behm DG, Muehlbauer T, Kibele A, Granacher U. Effects of Strength Training Using Unstable Surfaces on Strength, Power and Balance Performance Across the Lifespan: A Systematic Review and Meta-analysis. Sports Med. 2015 Dec;45(12):1645-69. doi: 10.1007/s40279-015-0384-x. PMID 26359066
- [Background] Bird ML, Hill KD, Fell JW. A randomized controlled study investigating static and dynamic balance in older adults after training with Pilates. Arch Phys Med Rehabil. 2012 Jan;93(1):43-9. doi: 10.1016/j.apmr.2011.08.005. Epub 2011 Oct 5. PMID 21975148
- [Background] Buldt AK, Levinger P, Murley GS, Menz HB, Nester CJ, Landorf KB. Foot posture is associated with kinematics of the foot during gait: A comparison of normal, planus and cavus feet. Gait Posture. 2015 Jun;42(1):42-8. doi: 10.1016/j.gaitpost.2015.03.004. Epub 2015 Mar 12. PMID 25819716
- [Background] Bullo V, Bergamin M, Gobbo S, Sieverdes JC, Zaccaria M, Neunhaeuserer D, Ermolao A. The effects of Pilates exercise training on physical fitness and wellbeing in the elderly: A systematic review for future exercise prescription. Prev Med. 2015 Jun;75:1-11. doi: 10.1016/j.ypmed.2015.03.002. Epub 2015 Mar 12. PMID 25773473
- [Background] Caravaggi P, Pataky T, Gunther M, Savage R, Crompton R. Dynamics of longitudinal arch support in relation to walking speed: contribution of the plantar aponeurosis. J Anat. 2010 Sep;217(3):254-61. doi: 10.1111/j.1469-7580.2010.01261.x. Epub 2010 Jul 14. PMID 20646107
- [Background] Casonatto J, Yamacita CM. Pilates exercise and postural balance in older adults: A systematic review and meta-analysis of randomized controlled trials. Complement Ther Med. 2020 Jan;48:102232. doi: 10.1016/j.ctim.2019.102232. Epub 2019 Nov 3. PMID 31987246
- [Background] Cote KP, Brunet ME, Gansneder BM, Shultz SJ. Effects of Pronated and Supinated Foot Postures on Static and Dynamic Postural Stability. J Athl Train. 2005 Mar;40(1):41-46. PMID 15902323
- [Background] Dingenen B, Malfait B, Nijs S, Peers KH, Vereecken S, Verschueren SM, Janssens L, Staes FF. Postural Stability During Single-Leg Stance: A Preliminary Evaluation of Noncontact Lower Extremity Injury Risk. J Orthop Sports Phys Ther. 2016 Aug;46(8):650-7. doi: 10.2519/jospt.2016.6278. Epub 2016 Jul 3. PMID 27374015
- [Background] Dlugosz-Bos M, Filar-Mierzwa K, Stawarz R, Scislowska-Czarnecka A, Jankowicz-Szymanska A, Bac A. Effect of Three Months Pilates Training on Balance and Fall Risk in Older Women. Int J Environ Res Public Health. 2021 Apr 1;18(7):3663. doi: 10.3390/ijerph18073663. PMID 33915843
- [Background] Domjanic J, Fieder M, Seidler H, Mitteroecker P. Geometric morphometric footprint analysis of young women. J Foot Ankle Res. 2013 Jul 25;6(1):27. doi: 10.1186/1757-1146-6-27. PMID 23886074
- [Background] Donatoni da Silva L, Shiel A, Sheahan J, McIntosh C. Six weeks of Pilates improved functional mobility, postural balance and spatiotemporal parameters of gait to decrease the risk of falls in healthy older adults. J Bodyw Mov Ther. 2022 Jan;29:1-9. doi: 10.1016/j.jbmt.2021.06.014. Epub 2021 Jun 23. PMID 35248255
- [Background] Ekstrom RA, Donatelli RA, Carp KC. Electromyographic analysis of core trunk, hip, and thigh muscles during 9 rehabilitation exercises. J Orthop Sports Phys Ther. 2007 Dec;37(12):754-62. doi: 10.2519/jospt.2007.2471. Epub 2007 Aug 29. PMID 18560185
- [Background] Elsayed W, Alotaibi S, Shaheen A, Farouk M, Farrag A. The combined effect of short foot exercises and orthosis in symptomatic flexible flatfoot: a randomized controlled trial. Eur J Phys Rehabil Med. 2023 Jun;59(3):396-405. doi: 10.23736/S1973-9087.23.07846-2. Epub 2023 Mar 29. PMID 36988565
- [Background] Farokhmanesh K, Shirzadian T, Mahboubi M, Shahri MN. Effect of foot hyperpronation on lumbar lordosis and thoracic kyphosis in standing position using 3-dimensional ultrasound-based motion analysis system. Glob J Health Sci. 2014 Jun 17;6(5):254-60. doi: 10.5539/gjhs.v6n5p254. PMID 25169004
- [Background] Flores DV, Mejia Gomez C, Fernandez Hernando M, Davis MA, Pathria MN. Adult Acquired Flatfoot Deformity: Anatomy, Biomechanics, Staging, and Imaging Findings. Radiographics. 2019 Sep-Oct;39(5):1437-1460. doi: 10.1148/rg.2019190046. PMID 31498747
- [Background] Ghasemi MS, Koohpayehzadeh J, Kadkhodaei H, Ehsani AA. The effect of foot hyperpronation on spine alignment in standing position. Med J Islam Repub Iran. 2016 Dec 28;30:466. eCollection 2016. PMID 28491841
- [Background] Giacomini MB, da Silva AM, Weber LM, Monteiro MB. The Pilates Method increases respiratory muscle strength and performance as well as abdominal muscle thickness. J Bodyw Mov Ther. 2016 Apr;20(2):258-64. doi: 10.1016/j.jbmt.2015.11.003. Epub 2015 Nov 10. PMID 27210841
- [Background] Hillstrom HJ, Song J, Kraszewski AP, Hafer JF, Mootanah R, Dufour AB, Chow BS, Deland JT 3rd. Foot type biomechanics part 1: structure and function of the asymptomatic foot. Gait Posture. 2013 Mar;37(3):445-51. doi: 10.1016/j.gaitpost.2012.09.007. Epub 2012 Oct 26. PMID 23107625
- [Background] Holowka NB, Lieberman DE. Rethinking the evolution of the human foot: insights from experimental research. J Exp Biol. 2018 Sep 6;221(Pt 17):jeb174425. doi: 10.1242/jeb.174425. PMID 30190415
- [Background] Huang C, Chen LY, Liao YH, Masodsai K, Lin YY. Effects of the Short-Foot Exercise on Foot Alignment and Muscle Hypertrophy in Flatfoot Individuals: A Meta-Analysis. Int J Environ Res Public Health. 2022 Sep 22;19(19):11994. doi: 10.3390/ijerph191911994. PMID 36231295
- [Background] Huang TH, Chou LW, Huang CY, Wei SW, Tsai YJ, Chen YJ. H-reflex in abductor hallucis and postural performance between flexible flatfoot and normal foot. Phys Ther Sport. 2019 May;37:27-33. doi: 10.1016/j.ptsp.2019.02.004. Epub 2019 Feb 19. PMID 30818085
- [Background] Ivanenko Y, Gurfinkel VS. Human Postural Control. Front Neurosci. 2018 Mar 20;12:171. doi: 10.3389/fnins.2018.00171. eCollection 2018. PMID 29615859